CLINICAL TRIAL: NCT05611918
Title: The Repeated Assessment of Survivors in ICH (REASSESS ICH)
Brief Title: REpeated ASSEssment of SurvivorS in Intracerebral Hemorrhage Study
Acronym: ICH03
Status: Enrolling by invitation | Type: Observational
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH); National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Other Study IDs: IRB00311985; R01NS120557 (NIH)
Record Dates: First submitted 2022-11-03; First posted 2022-11-10 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Intra Cerebral Hemorrhage; ICH - Intracerebral Hemorrhage; ICH; Hemorrhage; Stroke; Clot (Blood); Brain; Clot Blood; Cognitive Decline; Cognitive Impairment; Survivorship; Memory Impairment; Motor Activity
Keywords: Intracerebral hemorrhage; Stroke; Cognitive Impairment
MeSH Terms: conditions — Cerebral Hemorrhage; Hemorrhage; Stroke; Intracranial Thrombosis; Thrombosis; Cognitive Dysfunction; Memory Disorders; Motor Activity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Complete Blood Count, Ribonucleic Acid, Deoxyribonucleic Acid
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The investigators propose to perform serial detailed cognitive, motor, behavioral, and blood collection follow-up using longitudinal structured telephone interviews of an anticipated 350 ICH survivors enrolled in Minimally Invasive Surgery Plus Alteplase for Intracerebral Hemorrhage Evacuation (MISTIE) III and ENRICH trials to identify specific cognitive and motor impairment and to perform RNA sequencing to evaluate for evidence of chronic inflammation. The investigators' expected sample size in 2022 accounts for mortality attrition of 10%/year.

DETAILED DESCRIPTION:
The REASSESS study will conduct long-term cognitive, functional, and neuropsychiatric performance assessments to determine if evacuation of spontaneous intracerebral hemorrhage (ICH) reduces the risk of later cognitive decline in the ageing brain. This study will compare rates of cognitive decline under two treatment strategies for intracerebral hemorrhage: the use of minimally invasive surgery with two similar techniques as performed in the MISTIE III and ENRICH trials, and the current standard of care using data from controls in MISTIE III and ENRICH and comparative data from The Ethnic/Racial Variations of ICH (ERICH) study (U-01-NS067963) extended into the ERICH-Longitudinal study (R01-NS093870) which followed over 900 of ERICH cases with serial cognitive examinations.

ELIGIBILITY:
Inclusion Criteria:

* Participants in the study must be survivors enrolled in MISTIE III and ENRICH trials at end of each trial's final follow-up (day 365 in MISTIE III and day 180 in ENRICH). Relatives of known survivors that are found to be deceased since the end of each trial will be interviewed to capture relevant data.

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study populations includes all surviving cases identified and recruited through the 5-year durations of the MISTIE III and ENRICH trials and with follow-up periods extending from 2013-2017 and 2016-2022, respectively.
Sampling Method: Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2023-05-23 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
To determine if surgical clot reduction after ICH reduces the risk of progressive cognitive decline. | 24 months
  Primary outcome measure is the rate of cognitive decline which is based on a composite measure of global cognition using the National Institute on Aging Genetics Initiative for Late Onset Alzheimer Disease (NIA-LOAD) Battery.
  Clot reduction measure will be obtained from semi-automated computerized volumetrics using the OsiriX software.
  National Institute on Aging Genetics Initiative for Late Onset Alzheimer Disease (NIA-LOAD) Battery is a 7-measure cognitive testing battery to assess change in episodic, semantic, and working memory in community-dwelling older persons with broad ability levels.

SECONDARY OUTCOMES:
To determine if there is a long-term benefit in survival and functional outcome from minimally invasive surgery whether or not cognitive decline occurs | 24 months
  Survival and poor functional outcome (Modified Rankin Score (mRS) 4-6) will be calculated separately for cases with <=20 mL and >20 mL volume. We will use statistical modeling similar to Aim 1 to compute and calculate differences in hazard ratios for risk of mortality and poor outcome among <=20 mL and >20 mL survivors. We will assess interaction between cognitive decline and functional performance decline to evaluate whether these decline together.
  Secondary outcome measures include the following: Modified Rankin Scale score (mRS), NIH Stroke Scale (NIHSS), Motor Assessment Scale (MAS), Western Aphasia Battery (WAB), Mini Mental Status Exam (MMSE), Barthel Index (BI), De Jong Gierveld Loneliness Scale, EuroQol 5 Dimension (EQ-5D), Activities of Daily Living (ADL) and fall history, Telephone Interview for Cognitive Status (TICS), Informant Questionnaire on Cognitive Decline in the Elderly (IQ-CODE) and Center for Epidemiological Studies Depression (CES-D).

CONTACTS AND LOCATIONS:
Overall Officials: Wendy Ziai, MD, Principal Investigator — Johns Hopkins University
Locations (26):
- United States (26):
  - University of Alabama at Brimingham, Birmingham, Alabama
  - Scripps Health, La Jolla, California
  - Dignity Health component - St. Joseph's Hospital and Medical Center, Sacramento, California
  - Stanford University, Stanford, California
  - Yale University, New Haven, Connecticut
  - Mayo Clinic, Jacksonville, Jacksonville, Florida
  - CommonSpirit (formerly Mercy San Juan Medical Center; dignity health), Chicago, Illinois
  - University of Illinois at Chicago, Chicago, Illinois
  - University of Kansas Medical Center, Fairway, Kansas
  - University of Louisville, Louisville, Kentucky
  - University of Maryland Baltimore, Baltimore, Maryland
  - Johns Hopkins Hospital, Baltimore, Maryland
  - University of Michigan, Ann Arbor, Michigan
  - Henry Ford Health System, Detroit, Michigan
  - Hennepin Healthcare Research Institute, Minneapolis, Minnesota
  - Washington University in St. Louis, School of Medicine, St Louis, Missouri
  - Rutgers - Robert Wood Johnson Medical School, Piscataway, New Jersey
  - University of New Mexico, Albuquerque, New Mexico
  - Albert Einstein Montefiore, The Bronx, New York
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - University of Cincinnati, Cincinnati, Ohio
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - University of Texas, Houston Health Science Center, Houston, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Inova Health System Foundation, Fairfax, Virginia

IPD SHARING:
Plan to Share IPD: Yes
NIH policy states grant award recipients must make unique resources readily available for research purposes to qualified individuals within the scientific community after publication. Drs. Ziai and Flaherty are committed to sharing resources, products, and data generated in this study. They are aware of and agree to abide by the principles for sharing research resources as described by NIH in "Principles and Guidelines for Recipients of NIH Research Grants and Contracts on Obtaining and Disseminating Biomedical Research Programs."
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 9 months of database lock
Access Criteria: We will share individual-participant-level data, in a de-identified format in compliance with the HIPAA privacy rule, which will make the data free of identifiers that would permit linkages to the research participants and free of content that would create unacceptable risk of subject identification.

REFERENCES:
- [Derived] Ziai W, Woo D, Sansing L, Hanley D, Ostapkovich N, Triene K, Gilkerson LA, Thompson R, Walborn N, Lane K, McBee N, Langefeld CD, Howard TD, Vagal A, Flaherty ML. The REpeated ASSEssment of SurvivorS in intracerebral haemorrhage: protocol for a multicentre, prospective observational study. BMJ Open. 2025 Feb 6;15(2):e094322. doi: 10.1136/bmjopen-2024-094322. PMID 39915023